CLINICAL TRIAL: NCT04144881
Title: Angiographic Control Vs. Ischemia-driven Management of Patients Undergoing Percutaneous Revascularization of the Unprotected Left Main Coronary Artery with Second-generation Drug Eluting Stents: the PULSE Trial
Brief Title: Angiographic Control Vs. Ischemia-driven Management of Patients Treated with PCI on Left Main with Drug-eluting Stents
Acronym: PULSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Collaborators: Università degli Studi di Ferrara (Other); Ospedale San Luigi Gonzaga, Orbassano (Unknown); Ospedale Santa Croce-Carle Cuneo (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); AUSL Romagna Rimini (Other); University of Ferrara Department of Life Sciences and Biotechnology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PULSE-ULM
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Acute Coronary Syndrome; Stable Chronic Angina; Coronary Artery Disease; Left Main Coronary Artery Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Stable; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- coronary computed tomography (Experimental)
  Interventions: Diagnostic Test: coronary computed tomography
- conservative (ischemia-guided) management (No Intervention)

INTERVENTIONS:
Diagnostic Test: coronary computed tomography — patients randomized in this arm will perform computed coronary tomography 6 months after the index percutaneous revascularization on unprotected left main artery
  Arms: coronary computed tomography

SUMMARY:
The present study aims to compare a planned angiographic control (PAC) follow-up strategy vs. conservative management for patients treated with drug-eluting stents on unprotected left main artery in a prospective, randomized setting. PAC will be performed by coronary computed tomography (CCT), to avoid the limitations of the invasive coronary angiography which is usually employed to perform PAC. The superiority of a PAC-based approach will be tested on a hard clinical end-point such as the incidence of major adverse cardiovascular events. The investigators will also assess the performance of CCT as a tool to perform PAC.

DETAILED DESCRIPTION:
Given the undefined picture surrounding the appropriateness of planned angiographic control (PAC) following percutaneous coronary intervention (PCI) of the unprotected left main (ULM) with drug-eluting stents (DES), our aim is to evaluate, in a prospective, randomized, setting, the potential benefits of a PAC-based strategy vs. ischemia and symptoms driven conservative management. The disease of the native ULM is associated with an unfavorable prognostic outcome, which can be at least partially reversed by revascularization. Significant stenosis of the stented ULM caused by in-stent restenosis (ISR), however, presents some peculiar pathophysiological, flow-related and shear-stress features, which partly makes it a distinct disease as compared to native vessel atherosclerosis. Treatment of ISR, moreover, is a scarcely standardized and often complex procedure; some uncertainties still persist regarding the best strategy to treat ISR (stent-in-stent, drug-eluting balloons, dilation with conventional balloons). Computed coronary tomography (CCT) can precisely and not-invasively assess the presence of ISR in the stented ULM, without exposing the patients to the risks of invasive catheterization. CCT may provide an accurate reconstruction of the stented vessels, exposing the patients to a limited amount of contrast dye (approximately, 80-100 cc) and of radiation dose (approximately, 92 mGy). CCT has a very high negative predictive value for ISR, thus limiting the negative impact of the indiscriminate execution of invasive angiography on all patients treated by PCI of the ULM. Only patients with relevant ISR of ULM at CCT will undergo coronary angiography to confirm the presence of critical stenosis, and fractional flow reserve (FFR) and/or intravascular ultrasound (IVUS) will be performed in dubious cases.

An increased rate of PCI has to be taken in to account with a PAC-based approach. However, with the accurate, stepwise selection of the patients and the lesions amenable to PCI of our study protocol, based on CCT, coronary angiography and, where necessary, FFR/IVUS, the increased rate of PCI is not expected to bear a negative prognostic impact. Based on these premises, our hypothesis is that early, appropriate, detection of ULM ISR and its subsequent treatment may positively impact patients' survival and reduce the incidence of adverse cardiovascular events.

Specific aim 1:

Evaluation of the effectiveness and safety of a PAC-based approach to follow-up patients treated by PCI of the ULM with DES-II

Specific aim 2:

Assessment of the incidence of ISR in patients undergoing PCI of the ULM with DES-II and evaluation of the diagnostic accuracy of CCT in the evaluation of ISR in the stented ULM

Specific Aim 3:

Assessment of the prognostic implications and safety of the PCI of ISR of the ULM detected by PAC as compared to conservative management with revascularization driven by symptoms and ischemia.

For this purpose in this prospective, randomized controlled trial (RCT), patients will be enrolled following the index percutaneous revascularization of ULM with DES. Patients will be randomized in a 1:1 fashion to PAC-based management with CCT vs.

symptoms and ischemia driven conservative management.

ELIGIBILITY:
Inclusion Criteria:

Patients with ULM disease treated by PCI with DES-II with the following inclusion criteria:

* Age 18-85.
* Glomerular filtration rate > 30 ml/min Indication to percutaneous revascularization of ULM according to Syntax score (< 33) or, in dubious cases, after Heart Team evaluation

Exclusion Criteria:

* Cardiogenic shock
* Refusal or inability to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 18 months after the index revascularization
  composite and mutual exclusive end point including death, cardiovascular death, myocardial infarction (MI) (excluding periprocedural MI), unstable angina (UA), stent thrombosis

SECONDARY OUTCOMES:
Target lesion revascularization (TLR) | 18 months after the index revascularization
  target lesion revascularization including any TLR, any unplanned TLR and TLR driven by PAC
All cause death | within 18 months from the index revascularization
  death from any cause occurring during follow up
stent thrombosis | within 18 months from the index revascularization
  Any stent thrombosis (definite, probable or possible)
CV death | within 18 months from the index revascularization
  death from cardiovascular causes
Myocardial infarction | within 18 months from the index revascularization
  Myocardial infarction defined as non ST elevation acute coronary syndrome (NST-ACS) or ST elevation myocardial infarction (STEMI)

OTHER OUTCOMES:
AKI | 2 days after CCT in the experimental arm
  Acute kidney injury (AKI) following CCT will constitute safety end-point
Renal function impairment | 18 months after the index revascularization
  reduction of glomerular filtration rate of >24% or end-stage chronic kidney disease
Overall bleedings | 18 months after the index revascularization
  Any bleeding regardless of severity, defined according to Bleeding Academic Research Consortium (BARC) criteria
Major bleedings | 18 months after the index revascularization
  BARC bleedings type III-IV-V
procedural complications | Index hospitalization
  Procedural complications following each percutaneous coronary intervention (PCI): periprocedural MI defined, arterial access site complications, acute kidney injury

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio D'Ascenzo, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (3):
- Italy (3):
  - AOU Città della Salute e della Scienza di Torino, Torino, Italy
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara
  - Ospedale San Luigi Gonzaga, Orbassano, Orbassano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Authors/Task Force members; Windecker S, Kolh P, Alfonso F, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Head SJ, Juni P, Kappetein AP, Kastrati A, Knuuti J, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Sousa Uva M, Stefanini GG, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A. 2014 ESC/EACTS Guidelines on myocardial revascularization: The Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS)Developed with the special contribution of the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eur Heart J. 2014 Oct 1;35(37):2541-619. doi: 10.1093/eurheartj/ehu278. Epub 2014 Aug 29. No abstract available. PMID 25173339
- [Background] Sheiban I, Moretti C, D'Ascenzo F, Chieffo A, Taha S, Connor SO, Chandran S, de la Torre Hernandez JM, Chen S, Varbella F, Omede P, Iannaccone M, Meliga E, Kawamoto H, Montefusco A, Mervyn C, Garot P, Sin L, Gasparetto V, Abdirashid M, Cerrato E, Biondi Zoccai G, Gaita F, Escaned J, Hiddick Smith D, Lefevre T, Colombo A. Long-Term (>/=10 Years) Safety of Percutaneous Treatment of Unprotected Left Main Stenosis With Drug-Eluting Stents. Am J Cardiol. 2016 Jul 1;118(1):32-9. doi: 10.1016/j.amjcard.2016.04.007. Epub 2016 Apr 26. PMID 27209125
- [Background] Cassese S, Byrne RA, Schulz S, Hoppman P, Kreutzer J, Feuchtenberger A, Ibrahim T, Ott I, Fusaro M, Schunkert H, Laugwitz KL, Kastrati A. Prognostic role of restenosis in 10 004 patients undergoing routine control angiography after coronary stenting. Eur Heart J. 2015 Jan 7;36(2):94-9. doi: 10.1093/eurheartj/ehu383. Epub 2014 Oct 8. PMID 25298237
- [Background] Alfonso F, Byrne RA, Rivero F, Kastrati A. Current treatment of in-stent restenosis. J Am Coll Cardiol. 2014 Jun 24;63(24):2659-73. doi: 10.1016/j.jacc.2014.02.545. Epub 2014 Mar 13. PMID 24632282
- [Background] Stone GW, Parise H, Witzenbichler B, Kirtane A, Guagliumi G, Peruga JZ, Brodie BR, Dudek D, Mockel M, Lansky AJ, Mehran R. Selection criteria for drug-eluting versus bare-metal stents and the impact of routine angiographic follow-up: 2-year insights from the HORIZONS-AMI (Harmonizing Outcomes With Revascularization and Stents in Acute Myocardial Infarction) trial. J Am Coll Cardiol. 2010 Nov 2;56(19):1597-604. doi: 10.1016/j.jacc.2010.08.608. Epub 2010 Oct 1. PMID 20888162
- [Background] Uchida T, Popma J, Stone GW, Ellis SG, Turco MA, Ormiston JA, Muramatsu T, Nakamura M, Nanto S, Yokoi H, Baim DS. The clinical impact of routine angiographic follow-up in randomized trials of drug-eluting stents: a critical assessment of "oculostenotic" reintervention in patients with intermediate lesions. JACC Cardiovasc Interv. 2010 Apr;3(4):403-11. doi: 10.1016/j.jcin.2010.01.010. PMID 20398868
- [Background] Lee JY, Park DW, Kim YH, Yun SC, Kim WJ, Kang SJ, Lee SW, Lee CW, Park SW, Park SJ. Incidence, predictors, treatment, and long-term prognosis of patients with restenosis after drug-eluting stent implantation for unprotected left main coronary artery disease. J Am Coll Cardiol. 2011 Mar 22;57(12):1349-58. doi: 10.1016/j.jacc.2010.10.041. PMID 21414531
- [Background] Biondi-Zoccai GG, Giraudi E, Moretti C, Sciuto F, Omede P, Sillano D, Garrone P, Trevi GP, Sheiban I. Impact of routine angiographic follow-up after percutaneous coronary drug-eluting stenting for unprotected left main disease: the Turin Registry. Clin Res Cardiol. 2010 Apr;99(4):235-42. doi: 10.1007/s00392-009-0112-3. Epub 2010 Jan 3. PMID 20047051
- [Background] Valgimigli M, Chieffo A, Lefevre T, Colombo A, Morice MC, Serruys PW. Revisiting the incidence and temporal distribution of cardiac and sudden death in patients undergoing elective intervention for unprotected left main coronary artery stenosis in the drug eluting stent era. EuroIntervention. 2007 Feb;2(4):435-43. PMID 19755282
- [Background] Roura G, Gomez-Lara J, Ferreiro JL, Gomez-Hospital JA, Romaguera R, Teruel LM, Carreno E, Esplugas E, Alfonso F, Cequier A. Multislice CT for assessing in-stent dimensions after left main coronary artery stenting: a comparison with three dimensional intravascular ultrasound. Heart. 2013 Aug;99(15):1106-12. doi: 10.1136/heartjnl-2013-303679. Epub 2013 May 30. PMID 23723447
- [Background] Serruys PW, Morice MC, Kappetein AP, Colombo A, Holmes DR, Mack MJ, Stahle E, Feldman TE, van den Brand M, Bass EJ, Van Dyck N, Leadley K, Dawkins KD, Mohr FW; SYNTAX Investigators. Percutaneous coronary intervention versus coronary-artery bypass grafting for severe coronary artery disease. N Engl J Med. 2009 Mar 5;360(10):961-72. doi: 10.1056/NEJMoa0804626. Epub 2009 Feb 18. PMID 19228612
- [Background] Buchanan GL, Chieffo A, Bernelli C, Montorfano M, Carlino M, Latib A, Figini F, Giannini F, Durante A, Ielasi A, Castelli A, Colombo A. Two-year outcomes following unprotected left main stenting with first vs. new-generation drug-eluting stents: the FINE registry. EuroIntervention. 2013 Nov;9(7):809-16. doi: 10.4244/EIJV9I7A134. PMID 24280157
- [Background] Tonino PA, De Bruyne B, Pijls NH, Siebert U, Ikeno F, van' t Veer M, Klauss V, Manoharan G, Engstrom T, Oldroyd KG, Ver Lee PN, MacCarthy PA, Fearon WF; FAME Study Investigators. Fractional flow reserve versus angiography for guiding percutaneous coronary intervention. N Engl J Med. 2009 Jan 15;360(3):213-24. doi: 10.1056/NEJMoa0807611. PMID 19144937
- [Background] D'Ascenzo F, Barbero U, Cerrato E, Lipinski MJ, Omede P, Montefusco A, Taha S, Naganuma T, Reith S, Voros S, Latib A, Gonzalo N, Quadri G, Colombo A, Biondi-Zoccai G, Escaned J, Moretti C, Gaita F. Accuracy of intravascular ultrasound and optical coherence tomography in identifying functionally significant coronary stenosis according to vessel diameter: A meta-analysis of 2,581 patients and 2,807 lesions. Am Heart J. 2015 May;169(5):663-73. doi: 10.1016/j.ahj.2015.01.013. Epub 2015 Feb 21. PMID 25965714
- [Background] Hicks KA, Tcheng JE, Bozkurt B, Chaitman BR, Cutlip DE, Farb A, Fonarow GC, Jacobs JP, Jaff MR, Lichtman JH, Limacher MC, Mahaffey KW, Mehran R, Nissen SE, Smith EE, Targum SL. 2014 ACC/AHA Key Data Elements and Definitions for Cardiovascular Endpoint Events in Clinical Trials: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Data Standards (Writing Committee to Develop Cardiovascular Endpoints Data Standards). J Am Coll Cardiol. 2015 Jul 28;66(4):403-69. doi: 10.1016/j.jacc.2014.12.018. Epub 2014 Dec 29. No abstract available. PMID 25553722
- [Background] Mehta RL, Kellum JA, Shah SV, Molitoris BA, Ronco C, Warnock DG, Levin A; Acute Kidney Injury Network. Acute Kidney Injury Network: report of an initiative to improve outcomes in acute kidney injury. Crit Care. 2007;11(2):R31. doi: 10.1186/cc5713. PMID 17331245
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Mehran R, Dangas G, Abizaid AS, Mintz GS, Lansky AJ, Satler LF, Pichard AD, Kent KM, Stone GW, Leon MB. Angiographic patterns of in-stent restenosis: classification and implications for long-term outcome. Circulation. 1999 Nov 2;100(18):1872-8. doi: 10.1161/01.cir.100.18.1872. PMID 10545431
- [Background] D'Ascenzo F, Iannaccone M, Giordana F, Chieffo A, Connor SO, Napp LC, Chandran S, de la Torre Hernandez JM, Chen SL, Varbella F, Omede P, Taha S, Meliga E, Kawamoto H, Montefusco A, Chong M, Garot P, Sin L, Gasparetto V, Abdirashid M, Cerrato E, Biondi-Zoccai G, Gaita F, Escaned J, Hiddick Smith D, Lefevre T, Colombo A, Sheiban I, Moretti C. Provisional vs. two-stent technique for unprotected left main coronary artery disease after ten years follow up: A propensity matched analysis. Int J Cardiol. 2016 May 15;211:37-42. doi: 10.1016/j.ijcard.2016.02.136. Epub 2016 Mar 3. PMID 26970964
- [Derived] D'Ascenzo F, Cerrato E, De Filippo O, Gaido L, Franze A, Iannaccone M, Wanha W, Santarelli A, Guiducci V, Barbero U, Fernandez Pereira C, Gatti M, Tebaldi M, Giammaria M, Boccuzzi G, Wojakowski W, di Pietro G, Placido R, Gili S, Depaoli A, Biondi Zoccai G, Tomassini F, Bruno F, Zugna D, Faletti R, Biscaglia S, Caglioni S, Varbella F, de Ferrari GM, Campo G. Computed Tomography Angiography or Standard Care After Left Main PCI? J Am Coll Cardiol. 2025 Nov 11;86(19):1724-1734. doi: 10.1016/j.jacc.2025.07.060. Epub 2025 Aug 31. PMID 40886174
- [Derived] De Filippo O, Bianco M, Tebaldi M, Iannaccone M, Gaido L, Guiducci V, Santarelli A, Zaccaro L, Depaoli A, Vaudano P, Quadri G, Gagnor A, Boccuzzi G, Solitro F, Cortese G, Guarnaccia C, Tore D, Veltri A, Franchin L, Angelini F, Garbo R, Giammaria M, Varbella F, Marchisio F, Fonio P, De Ferrari GM, Cerrato E, Campo G, D'Ascenzo F. Angiographic control versus ischaemia-driven management of patients undergoing percutaneous revascularisation of the unprotected left main coronary artery with second-generation drug-eluting stents: rationale and design of the PULSE trial. Open Heart. 2020 Oct;7(2):e001253. doi: 10.1136/openhrt-2020-001253. PMID 33122421